CLINICAL TRIAL: NCT07260955
Title: Effects of a Multimodal Telerehabilitation Program in Patients With Chronic Non-Specific Neck Pain: Randomized Clinical Trial.
Brief Title: Effects of a Multimodal Telerehabilitation Program in Patients With Chronic Non-Specific Neck Pain.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Daniel Pantaleón Hernández, Associate Teacher in Physiotherapy, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FIS-2024-009
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Chronic Neck Pain; Non-specific Neck Pain
Keywords: Neck muscles; Chronic neck pain; Telerehabilitation; Exercise therapy; Pain education
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: This will be a randomized controlled trial with 2 different groups.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Thoracic spine mobility, deep cervical flexor and extensor muscles strength training, thoracic muscles strength training and pain education through telerehabilitation.
  Interventions: Other: Thoracic and neck specific exercise program and education
- Control group (Active Comparator): Thoracic spine mobility, thoracic muscles strength training and pain education through telerehabilitation.
  Interventions: Other: Thoracic exercise program and education

INTERVENTIONS:
Other: Thoracic exercise program and education — Thoracic spine mobility, thoracic muscles strength training and pain education through telerehabilitation.
  Arms: Control group
Other: Thoracic and neck specific exercise program and education — Thoracic spine mobility, deep cervical flexor and extensor muscles strength training, thoracic muscles strength training and pain education through telerehabilitation.
  Arms: Experimental group

SUMMARY:
The purpose of this study is to evaluate the clinical results in pain intensity, neck disability, range of motion, endurance deep cervical muscles, forward head position and kinesiophobia through thoracic spine mobility, deep neck muscles and thoracic strength training and pain education protocol versus a thoracic spine mobility, thoracic strength training and pain education protocol in patients with chronic non-specific neck pain.

DETAILED DESCRIPTION:
The cervical spine is the most mobile region of the spine and must be strong enough to support the weight of the skull and thoracic spine is the most stiff region. In addition, patients often catastrophize their pain, it has a major impact on quality of life. Strength deficits of the deep cervical muscles are related to different clinical conditions, such as non-specific neck pain. Training and education protocols can help to improve pain, function, posture and cross-sectional area. However, there are no multimodal protocols in subjects with chronic non-specific neck pain including deep neck extensor and flexor muscles, thoracic spine mobility and pain education.

ELIGIBILITY:
Inclusion Criteria:

* Non-specific neck pain for at least the last 12 weeks.
* Pain intensity equal to or greater than 4 on the visual analog scale (VAS).
* Mild-moderate disability in the Neck Disability Index.
* Not reaching phase 2 in Craniocervical flexion test.
* Availability and skill to do video calls.
* Understanding Spanish.

Exclusion Criteria:

* Other type of neck pain.
* Previous neck surgery.
* Diagnosed metabolic diseases.
* Red flags (infection, tumors, rheumatic arthritis, or cardiovascular disease).
* History of cardio-respiratory disease that contraindicates high-intensity exercise.
* Fibromyalgia
* Pregnancy
* Physiotherapeuthic treatment continued in the last 3 month.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Baseline, 6 weeks, 1 month follow-up
  Measured by Visual Analogue Scale.
Neck Disability | Baseline, 6 weeks, 1 month follow-up
  Measured by the Spanish version of Neck Disability Index Questionnaire.

SECONDARY OUTCOMES:
Activation of deep neck flexors muscles. | Baseline, 6 weeks, 1 month follow-up
  Measured by Cranio-cervical flexion test
Forward head posture | Baseline, 6 weeks, 1 month follow-up
  Measured by craniovertebral angle.
Cervical range of motion | Baseline, 6 weeks, 1 month follow-up
  Measured by CROM(Cervical Range-of-Motion Instrument). Cervical flexion, extension, right/left side bending and right/left rotation.
Kinesiophobia | Baseline, 6 weeks, 1 month follow-up
  Measured with Spanish version of Tampa Scale
Global Rating of Change | 1 month follow-up
  Measured by Global Rating of Change Scale

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pantaleon-Hernandez, Principal Investigator — Universitat Internacional de Cataluña
Locations (1):
- Universitat Internacional de Cataluña, Sant Cugat del Vallès, Spain